CLINICAL TRIAL: NCT05185336
Title: Ultrasound Assessment of Gastric Volume and Aspiration Risk Evaluation in the Fasted Pediatric Cerebral Palsy Patients.
Brief Title: Ultrasound Assessed Gastric Volume in the Fasted Pediatric Cerebral Palsy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B-2104-681-301
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: ultrasound assessment — gastric volume assessment by ultrasound

SUMMARY:
In patients with cerebral palsy, delayed gastric emptying and esophageal sphincter dysfunction are very commonly observed.

Pulmonary aspiration of gastric contents causes aspiration pneumonia, which greatly affects patients' prognosis, including hospital stay and mortality.

In the case of patients with cerebral palsy, there is a limitation in respiratory function, so more attention is required.

Therefore, this study aims to evaluate the risk of aspiration by measuring gastric volume after fasting for surgery in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* patients with cerebral palsy under the age of 18 scheduled surgery under general anesthesia

Exclusion Criteria:

* the patient who feed through Levin tube or gastrostomy tube
* refusal to participate

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with cerebral palsy under the age of 18 scheduled surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
gastric volume | preoperative 20 minutes
  -7.8 + (3.5 x RLD CSA) + 0.127 X age (months)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea